CLINICAL TRIAL: NCT02544919
Title: Impact of Pretreatment With Omega 3 Enriched Lipid Emulsion on Early Neurological Complications After Living Donor Liver Transplantation. A Randomized Controlled Trial>
Brief Title: Lipids and Neurological Complications in Liver Transplantation
Acronym: LNCLT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Yassen, Professor of Anesthesia and Intensive care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SMOF_NEURO_1
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2016-07

CONDITIONS: Neurological Complications
Keywords: SMOF; neurological complications; neurotoxicity; liver transplantation; Lipid emulsions
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — SMOFlipid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): No Intervention group: Patients do not receive any lipid emulsion of any type during the study period
- SMOF Group (Active Comparator): Intervention Group: Patients receive 1 gm.kg.day-1 SMOFlipid for 48 hours before the operation and 5 days post-operatively.
  Interventions: Drug: SMOF lipid (SMOFLIPID) pre treatment

INTERVENTIONS:
Drug: SMOF lipid (SMOFLIPID) pre treatment — Experimental Arm
  Other Names: Experimental group
  Arms: SMOF Group

SUMMARY:
To study the impact of pretreatment of living donor liver transplantation recipients with SMOF lipid on the incidence and severity of post-transplantation neurological complications in patients receiving tacrolimus based immunosuppression protocol

DETAILED DESCRIPTION:
All patients included in the study will receive the same immuno-suppression protocol based on tacrolimus and mycophenolate mofetil after the induction immuno-suppression during the intra-operative period.

Patients will have a full history taking and full neurological examination 48 hours prior to the designated operative date as a basal record.

the control group will not receive any lipid infusions at all the treatment group will receive the study emulsion (SMOF lipid 20% - Fresenius Kabi) starting 48 hours before the planned surgery day and will continue to receive it for 5 post-operative days by intravenous infusion.

During the post-operative period. patients will be assessed daily by full neurological examination as will as patient complaints (symptoms) related to neurological status for diagnosis of any neurological conditions (complications) that might arise during the study period.

Data will be analysed compared to the basal value in each group and between both control and intervention groups using the appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Adult living donor liver transplant recipients of either sex

Exclusion Criteria:

* MELD score > 30
* Retransplantation
* Budd Chiari syndrome
* Diabetes more than 10 years

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
post-transplant neurological complications | 5 post-operative days
  Number of participants who develop neurological complications

SECONDARY OUTCOMES:
Graft functions | 5 post-operative days
  the laboratory parameters for graft functions in both groups
survival | 30 days
  one month mortality

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Yassen, MD, Principal Investigator — MAnsoura Faculty of Medicine
Locations (1):
- Liver transplantation project - Gastroenterology surgical center - Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt